CLINICAL TRIAL: NCT02771587
Title: Effects of Alcohol and Energy Drinks on Driving Performance and Bleeding Risk
Brief Title: Interaction of Alcohol With Energy Drinks
Acronym: AEDED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Clara Pérez, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: IMIMFTCL/AEDED
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol-Related Disorders; Drinking and Driving
Keywords: alcohol; energy drink; coagulability; caffeine; taurine; driving performance
MeSH Terms: conditions — Alcohol-Related Disorders; Driving Under the Influence | interventions — Ethanol; Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Alcohol and energy drink (Experimental): Alcohol 60 g, multiple dose (30 g+30 g), oral administration. 3 energy drinks (750 ml), multiple dose (375 ml+375 ml), oral administration.
  Interventions: Dietary Supplement: Alcohol and energy drink
- Alcohol (Active Comparator): Alcohol 60 g, multiple dose (30 g+30 g), oral administration. 3 non-caffeinated soft drinks (750 ml), multiple dose (375 ml+375 ml), oral administration.
  Interventions: Dietary Supplement: Alcohol
- Energy drink (Active Comparator): 3 energy drinks (750 ml), multiple dose (375 ml+ 375 ml), oral administration. Font Vella water (188ml), multiple dose (94 ml+ 94 ml), oral administration.
  Interventions: Dietary Supplement: Energy drink
- Placebo (Placebo Comparator): 3 non-caffeinated soft drinks (750 ml), multiple dose (375 ml+375 ml), oral administration.
  Font Vella water (188ml), multiple dose (94 ml+ 94 ml), oral administration.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alcohol and energy drink — Multiple oral dose of alcohol Multiple oral dose of energy drink
  Arms: Alcohol and energy drink
Dietary Supplement: Alcohol — Multiple oral dose of alcohol
  Arms: Alcohol
Dietary Supplement: Energy drink — Multiple oral dose of energy drink
  Arms: Energy drink
Dietary Supplement: Placebo — Multiple oral dose of water Multiple oral dose of non-caffeinated soft drink
  Other Names: Non-active treatment
  Arms: Placebo

SUMMARY:
The main objective of the project is to assess whether there is an interaction between the effects of ethanol and energy drinks on driving performance.

Secondary objectives include: to evaluate subjective effects (drunkenness) after administration of alcohol and energy drinks, to assess pharmacokinetics of alcohol, caffeine and taurine after alcohol and energy drinks administration and to assess if there is an increased risk of bleeding when both drinks are taken together.

DETAILED DESCRIPTION:
Consumption of energy drinks improve psychomotor performance and alertness. These drinks contain mostly caffeine, taurine and vitamins. Its consumption associated with ethanol may reduce feelings of drunkenness as the stimulant effects of caffeine could counteract the depressing effects of ethanol on the central nervous system. Reducing the perception of intoxication may predispose the intoxicated person to engage in risky behaviors such as driving under the influence of ethanol and therefore can increase the risk of a traffic accident. Furthermore, the combination of both beverages may increase the risk of bleeding in case of injury as anticoagulant effects have been described for ethanol while antiplatelet effects have been described for caffeine and taurine. A randomized clinical trial will be performed in healthy volunteers administering 4 treatment conditions: alcohol+energy drink, alcohol+placebo of energy drink, placebo of alcohol+energy drink and placebo of alcohol+placebo of energy drink. A multiple dose will be administered separated by 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Understand and accept the study's procedures and sign an informed consent form
* No evidence of somatic or psychiatric disorders as per past medical history and physical examination
* EKG, blood and urine tests taken before entry into the study within the normal range. Minor and transient abnormalities may be acceptable if, according to the Principal Investigator's criterion and the state of the art, they are felt to have no clinical relevance, entail no danger to the participant, and don't interfere with the product's assessment. These abnormalities and their non-relevance must be specifically justified in writing)
* Body mass index (BMI=weight/heigth2) between 19 and 27 kg/m2, weight between 50 and 100 kg
* For premenopausal females, a regular menstrual cycle of 26-32 days duration.
* Social or recreational alcohol consumption of at least 1 unit per day (or its equivalent [7 units] over the whole week) and having experienced drunkenness several times
* Regular consumption of beverages containing methylxanthines (at least 5 per week)
* Consumption of energy drinks several times previously
* Having a driving license

Exclusion Criteria:

* Evidence of a preexisting condition (including gastrointestinal, liver, or kidney disorders) that may alter the absorption, distribution, metabolism or excretion of the drug or symptoms suggestive of drug-induced gastrointestinal irritation
* Previous psychiatric disorders, alcoholism, abuse of prescription drugs or illegal substances or regular consumption of psychoactive drugs
* Having donated blood or having participated in this same study in the preceding 8 weeks, or having participated in any clinical trial with drugs in the preceding 12 weeks
* Having had any somatic disease or having undergone major surgery in the 3 months prior to inclusion in the trial
* Individuals intolerant or having experienced a severe adverse reaction to alcohol or energy drinks
* Having regularly taken medication in the month before the trial, except for vitamins, herb-based remedies, dietary supplements that if, according to the Principal Investigator or his appointed collaborators' opinion, they pose no threat to the subjects and they won't interfere with the study's objectives. Single doses of symptomatic drugs taken during the week before the experimental session will not constitute an exclusion criterion if it can be assumed that it has been completely eliminated on the day of the experimental session
* Smokers of >5 cigarettes/day
* Consumption of >20 g/day of alcohol (females) or of >40 g/day (males)
* Daily consumption of more than 5 coffees, teas, cola drinks or other stimulant or xanthine-containing beverages in the 3 months prior to inclusion in the study
* Hepatitis B, hepatitis C or human immunodeficiency virus-positive individuals
* Pregnant or lactating women, or those using hormonal or unreliable contraceptive methods during the study period. Complete abstinence, intrauterine devices, double barrier methods or a vasectomized sexual partner will be considered acceptable
* Women with amenorrhea or suffering severe premenstrual syndrome
* Individuals of Asian ascent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in tracking test performance | From baseline till 4 hours after administration
  The total time outside the road will be measured in the tracking test

SECONDARY OUTCOMES:
Change in simple reaction time (SRT) | From baseline till 4 hours after administration
  Test will be performed using the computerized cognitive testing battery CANTAB and mean latency will be measured
Change in movement estimation | From baseline till 4 hours after administration
  The lapse of time between actual and predicted time will be measured in a movement estimation task
Change in memory function | From baseline till 4 hours after administration
  The N-Back test will be performed with 2 different options: 0 back test and 2 back test
Change in drunkenness | From baseline till 8 hours after administration
  Drunkenness will be measured using a visual analog scale (0-100 mm)
Change in drowsiness | From baseline till 8 hours after administration
  Drowsiness will be measured using a visual analog scale (0-100 mm)
Change in headache | From baseline till 8 hours after administration
  Headache will be measured using a visual analog scale (0-100 mm)
Change in palpitations | From baseline till 8 hours after administration
  Palpitations will be measured using a visual analog scale (0-100 mm)
Change in anxiety | From baseline till 8 hours after administration
  Anxiety will be measured using a visual analog scale (0-100 mm)
Change in subjective effects measured with Addiction Research Center Inventory (ARCI) | From baseline till 8 hours after administration
  Subjective effects of alcohol and caffeine will be measured using Addiction Research Center Inventory
Change in subjective effects measured with Biphasic alcohol effects scale (BAES) | From baseline till 8 hours after administration
  Subjective effects of alcohol will be measured using BAES
Change in blood pressure | From baseline till 8 hours after administration
  Systolic and diastolic blood pressure will be measured
Change in heart rate | From baseline till 8 hours after administration
  Heart rate will be measured
Change in oral temperature | From baseline till 8 hours after administration
  Oral temperature will be measured
Number of participants with serious and non-serious adverse events | From inclusion till one week after the last experimental session
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators
Area under the concentration-time curve (AUC 0-8h) of ethanol blood concentrations | From baseline till 8 hours after administration
  Calculation of AUC of ethanol concentrations obtained baseline and 0.25, 0.50h , 0.75, 1, 1.50, 1.75, 2, 2.25, 2.5, 3, 4, 6 and 8h after administration
Area under the concentration-time curve (AUC 0-8h) of taurine blood concentrations | From baseline till 8 hours after administration
  Calculation of AUC of ethanol concentrations obtained baseline and 0.50,1, 1.50, 2, 4, 6 and 8h after administration
Area under the concentration-time curve (AUC 0-8h) of caffeine blood concentrations | From baseline till 8 hours after administration
  Calculation of AUC of ethanol concentrations obtained baseline and 0,25, 0.50,1, 1.50, 2, 3, 4, 6 and 8h after administration
Area under the concentration-time curve (AUC 0-8h) of ethanol breath air concentrations | From baseline till 8 hours after administration
  Calculation of AUC of ethanol concentrations obtained baseline and 0.25, 0.50, 0.75,1, 1.50, 1.75, 2, 2.25, 2.5, 3, 4, 6 and 8h after administration
Maximum concentration (Cmax) of taurine | From baseline till 8 hours after administration
Maximum concentration (Cmax) of ethanol | From baseline till 8 hours after administration
Maximum concentration (Cmax) of caffeine | From baseline till 8 hours after administration
Time to reach maximum concentration (tmax) of ethanol | From baseline till 8 hours after administration
Time to reach maximum concentration (tmax) of caffeine | From baseline till 8 hours after administration
Time to reach maximum concentration (tmax) of taurine | From baseline till 8 hours after administration
Blood coagulation prothrombin | From baseline till 2 hours after administration
  Prothrombin time (PT) and ratio will be measured
Blood coagulation thromboplastin | From baseline till 2 hours after administration
  Activated partial thromboplastin time (APTT) and ratio will be measured
Platelet aggregation (function) | From baseline till 2 hours after administration
  Platelet function (PFA) will be measured
Platelet count | From baseline till 2 hours after administration
  Platelet count will be measured
Change in willingness to drive | From baseline till 6 hours after administration
  Willingness to drive in 3 different situations will be measured by means of a visual analog scale
Like the drug (drink) | At the end of each experimental session
  Drug liking will be measured using a visual analog scale (0-100 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Pérez Mañá, PhD, MD, Principal Investigator — IMIM
Locations (2):
- Spain (2):
  - IMIM, Barcelona, Barcelona
  - Parc de Salut Mar-IMIM, Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Mana C, Mateus JA, Diaz-Pellicer P, Diaz-Baggerman A, Perez M, Pujadas M, Fonseca F, Papaseit E, Pujol J, Langohr K, de la Torre R. Effects of Mixing Energy Drinks With Alcohol on Driving-Related Skills. Int J Neuropsychopharmacol. 2022 Jan 12;25(1):13-25. doi: 10.1093/ijnp/pyab051. PMID 34338762